CLINICAL TRIAL: NCT05344625
Title: Ketamine-Assisted Psychotherapy Viability in Treating Cancer-Related Emotional Distress
Acronym: KAPTIVATED
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study team is not moving forward with protocol
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0418
Record Dates: First submitted 2022-03-31; First posted 2022-04-25 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cancer-related Problem/Condition; Depressive Symptoms; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine Assisted Psychotherapy (Experimental): 3 KAP sessions lasting approximately 3 hours using less than or equal to 60mg or 1mg/kg of intramuscular Ketalar as the facilitating chemical. KAP sessions will be supplemented with integration sessions occurring the following day and 1 month after the final KAP session.
  Interventions: Drug: Ketamine 100 MG/ML

INTERVENTIONS:
Drug: Ketamine 100 MG/ML — Ketamine Assisted Psychotherapy

SUMMARY:
The present study will investigate if ketamine-assisted psychotherapy during palliative radiation therapy is safe, feasible, and effective at reducing psychological distress.

DETAILED DESCRIPTION:
Patients prescribed palliative radiation therapy with moderate-severe cancer-related anxiety or depression will be prescribed 3 Ketamine Assisted Psychotherapy (KAP) sessions. At the time of enrollment, they will complete surveys to assess depression, anxiety, and existential distress. KAP will be preceded by a preparatory session during which the subjects will virtually meet their the KAP clinical team, discuss important stressors or concerns, and prepare for KAP. Each KAP session will last approximately 3 hours during which patients will receive an individualized dose of Ketalar intramuscularly, and after the ketamine experience subsides, the patient will discuss the experience with a psychotherapist trained in KAP. A virtual integration session will occur the day after each KAP session as it provides patients with an opportunity to work collaboratively with their assigned therapist in a manner that can help translate any insights from their preparation and KAP sessions into actionable goals. Depression, anxiety, and existential distress will be measured throughout the trial to assess the impact from KAP.

ELIGIBILITY:
Inclusion Criteria:

* Subject have provided informed consent
* Male or female ≥ 21 to ≤ 65years of age at signing of informed consent
* Moderate-severe anxiety or depression related to cancer as measured by the GRID-HAM-D17 (depression) or the HAM-A (anxiety)
* Prescribed a radiation therapy course with palliative intent. Radiation therapy will be given priority with respect to scheduling and delivery over appointments related to KAP. Patients may begin the KAP process as soon as they are able after enrollment as long as it does not interfere with or delay receipt of radiation therapy. The timing of KAP/ RT can be either concurrent or sequential with RT coming first based on convenience to the patient and treatment teams, although completing the treatment expediently will be encouraged. Total treatment package time should be less than 3 months from CT simulation.
* A female subject of childbearing potential who is sexually active with a non-sterilized male partner must agree to consistently and correctly use a highly effective method of contraception with a failure rate of < 1% per year (Appendix 1) during the study and for at least 90 days after study drug administration. If a hormonal contraceptive is used, it must have been initiated at least 1 month before dosing.
* Negative pregnancy test (women only)
* Female subject of non-childbearing potential must be either: surgically sterile (hysterectomy, tubal ligation, or bilateral oophorectomy), or post-menopausal with amenorrhea for at least 2 years and documented follicle-stimulating hormone (FSH) levels ≥30 mIU/mL, or mL or must use a medically accepted double-barrier contraceptive method during the study and for at least 90 days after study drug administration.
* Male subject must agree to use prophylactic contraception
* Patients receiving chemotherapy, hormonal therapy, radiation therapy, biologic therapies may participate while receiving those therapies. Continuing hormonal therapy, chemotherapy, or radiation treatment is acceptable if the patient is tolerating the therapy or treatment in a sufficient fashion to allow administration of intramuscular ketamine
* Agree that for one week preceding each KAP session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the research team. Exceptions will be evaluated by the research team and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals
* Agree not to use nicotine for at least 2 hours before KAP administration, and not again until questionnaires have been completed approximately 7 hours after KAP administration.
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of KAP session days. If the patient does not routinely consume caffeinated beverages, he or she must agree not to do so on KAP session days.
* Agree not to take any PRN medications on the mornings of KAP sessions, with the exception of daily opioid pain medication. Non-routine PRN medications for treating breakthrough pain that were taken in the 24 hours before the KAP session may result in rescheduling the treatment session, with the decision at the discretion of the investigators.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each KAP administration. As described elsewhere, exceptions include daily use of caffeine, nicotine, and opioid pain medication.
* Willingness to not driving for 24 hours following study drug administration
* English proficiency
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Karnofsky Performance Scale (KPS) index of 60 or less
* Patients will be excluded if they are in treatment in another clinical trial involving an investigational product for treatment of cancer.
* Hepatic dysfunction as indicated by the following values:

  * -- GGT > 3 x ULN (upper limit of norm)
  * -- AST > 3 x ULN
  * -- ALT > 3 x ULN
  * -- Tot Bili > 3.0 mg/dl
* Known paraneoplastic syndrome or "ectopic" hormone production by the primary tumor such as the patient could have or be at risk for hypercalcemia, Cushing's syndrome, hypoglycemia, syndrome of inappropriate antidiuretic hormone secretion, or carcinoid syndrome
* Cardiovascular conditions: uncontrolled hypertension, angina, a clinically significant ECG abnormality (e.g. atrial fibrilation), TIA in the last 6 months, stroke, peripheral or pulmonary vascular disease (no active claudication)
* Systolic blood pressure >140mmHG or < 85 mmHg or diastolic blood pressure >90mmHg or heart rate of > 110 beat per minutes. Pulse oximetry of 94% or less.
* Epilepsy with history of seizures
* Renal insufficiency (creatinine clearance < 40 ml/min using the Cockraft and Gault equation)
* Uncontrolled hyperthyroidism (low thyroid stimulating hormone with high T3 or T4)
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Opioid pain medications (e.g. oxycodone sustained release, morphine sustained release -- which are usually taken at 12 hour intervals) will be allowed if the last dose occurred at least 12 hours before KAP administration; such medication will not be taken again until at least 6 hours after KAP administration.
* Current or history of schizophrenia, psychotic disorder, bipolar disorder, delusional disorder, paranoid personality disorder, substance use disorder, schizoaffective disorder, or borderline personality disorder, as assessed by medical history. Patients who have bipolar disorder but are not currently in a manic state may be included based on judgement of investigators.
* Patients with first or second-degree relatives with schizophrenia, non-substance induced psychotic disorder, or bipolar disorder
* Increased risk of intracranial pressure:

  * Recent ischemic or hemorrhagic cerebral vascular accident in the last 1 month.
  * Brain tumors with symptoms and signs of increased intracranial pressure.
  * Seizure in the last 6 months.
  * Head trauma with symptoms of increased intracranial pressure.
  * Hydrocephalus.
  * Uncontrolled nausea/vomiting/headache or ≥ grade 3 nausea despite one line of antiemetics
  * Recent traumatic brain injury
* Potential for adverse drug-drug interactions. Concomitant medications with significant potential to interact with study medications will be exclusionary if they cannot be tapered. These include the following:
* Regular benzodiazepine usage greater than 0.5mg of clonazepam/day or equivalent which cannot be stopped 1 day prior to ketamine injection
* Lamotrigine usage
* Usage of methylphenidate, phenobarbital, or amphetamine drugs within 5 half-lives of KAP
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ketamine or ketamine sensitivity
* Severe depression/anxiety which warrants immediate treatment with antidepressant or anxiolytic medication due to suicidal ideation
* History of alcoholism or drinking more than an average of 2 alcoholic beverage per day within past 5 years
* Female subject of childbearing potential who is not willing to use effective methods of birth controls or practice sexual abstinence up to 10 days following the last administration of ketamine.
* A positive pregnancy test at Screening
* History or evidence of any other clinically significant disorder, condition, or disease that in the opinion of the investigator or based on psychotherapist opinion would pose a risk to the subject safety or interfere with the study evaluation, procedure, or completion.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of population completing at least one KAP session. | Within 6 months from completion of radiation therapy
  The percentage of subjects who complete at least 1 session of KAP will be calculated, along with the associated 95% exact binomial confidence interval. The null hypothesis will be rejective if >50% of patients complete at least 1 KAP session.

SECONDARY OUTCOMES:
Depression and Anxiety | Within 6 months from completion of radiation therapy
  GRID-HAM-D-17 for depression and the HAM-A for anxiety. These forms will be completed at baseline (time of enrollment), at the completion of the ketamine psychotherapy sessions, and at the completion of consolidative psychotherapy. A subject will be considered a responder if they have a 50% decrease from baseline in GRID-HAM-D-17 score for depression and a 50% decrease in HAM-A score for anxiety. At each timepoint subsequent to baseline, the percentage of subjects who are responders will be calculated, along with the associated 95% exact binomial confidence interval. If feasible, a subset analysis will be carried out for patients with GRID-HAM-D-17 scores of at least 22 or HAM-A scores at least 25 at baseline.
Death and Dying Distress Scale (DADDS) | Within 6 months from completion of radiation therapy
  The change from baseline in DADDS will be calculated at each timepoint subsequent to baseline, and summarized by calculating the median change, along with the first and third quartiles, and the minimum and maximum.
Mystical Experience Questionnaire (MEQ-30) | Within 6 months from completion of radiation therapy
  The MEQ-30 will be assessed after every KAP session, and summarized by calculating the median, along with the first and third quartiles, and the minimum and maximum. These values will be compared to historical controls in the psilocybin population for reference.

IPD SHARING:
Plan to Share IPD: No